CLINICAL TRIAL: NCT03099811
Title: Contingency Management for Controlling Secondhand Smoke Exposures Among Asthmatic Children
Brief Title: Financial Incentives to Reduce Pediatric Tobacco Smoke Exposures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00064875
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Asthma; Incentives; Tobacco Smoking
MeSH Terms: conditions — Asthma; Tobacco Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Financial incentives + Smoking cessation program (Experimental): Caregiver and a social network member will receive financial incentives, in additional to enrollment in a state-sponsored smoking cessation program, based on nicotine biomarker measurements.
  Interventions: Behavioral: Incentive plan; Behavioral: Smoking cessation
- Intervention: Smoking cessation program (Other): Caregiver and a social network member will be enrolled in a state-sponsored smoking cessation program.
  Interventions: Behavioral: Smoking cessation

INTERVENTIONS:
Behavioral: Incentive plan — The caregiver and designated social network member can each receive monthly financial incentives over the 6 month time interval. Additional monthly incentives will be received at 3- and 6-months if the participant's previous two monthly biomarker levels were below the lower-limit cutoff.
  Other Names: Contingency management
  Arms: Intervention: Financial incentives + Smoking cessation program
Behavioral: Smoking cessation — Participants who wish to quit smoking will be referred upon study recruitment to the smoking cessation program that is provided at no-cost by the Maryland Department of Health and Mental Hygiene (DMMH). The DMMH provides standard counseling and nicotine replacement pharmacotherapies for clients and is offered online or at six health centers throughout Baltimore City.
  Other Names: Tobacco cessation

SUMMARY:
Secondhand smoke exposure (SHSe) is one of the most common and potentially modifiable environmental triggers for asthma. Financial incentivization may serve as an effective modality to reduce SHSe among pediatric asthmatics with potential down-stream benefits on improved asthma control and subsequent reduced healthcare utilization. This study plans on testing the feasibility and effectiveness of financial incentives to decrease SHSe, derived from primary caregivers and a member of their social network, of children with persistent asthma.

DETAILED DESCRIPTION:
The impact of continued cigarette usage is profoundly felt not only upon the primary smoker, but also among children where SHSe is linked with asthma exacerbations. Children with caregivers who are active smokers are more likely to utilize acute healthcare resources and miss more days of school due to asthma symptoms. Issues of pediatric smoke exposure are notably higher among low-income populations. This particular group has a greater amount of financial strain that increases their desire to cease smoking but is among the least successful at accomplishing this task. Aggressive marketing campaigns by cigarette companies have specifically targeted the urban poor but similar techniques by public health officials, though on a much diminished scale, have yet to completely counter the hold that this addictive product has on members of lower socioeconomic status. One approach that has demonstrated efficacy in reducing smoking in resistant populations emphasizes financial incentives. Incentives may provide a substitute for the gratification derived from nicotine if they are properly structured. This proposal applies a contingency management schema among caregivers of pediatric asthmatics and a member of their caregiver's social network - both of whom are likely major contributors to the child's total secondhand smoke exposure. A pilot two-arm randomized-control trial will be employed over a 6-month time interval.The study population will consist of the primary caregiver and a selected member of their social network, both of who are known active smokers, and contemplating smoking cessation; both individuals spend time (either indoors or outdoors) with the asthmatic child. We will recruit 50 caregiver-child-social network triads among a population of children diagnosed with uncontrolled, persistent asthma and routinely exposed to high levels of SHSe. Caregivers and members of their social network who are both active smokers will be randomized to receive standard smoking cessation strategies (n=25 triads) with or without financial incentives (n=25 triads). SHSe will be measured directly using salivary cotinine levels from children and home air nicotine levels. Caregiver and social network member smoking behaviors will be measured by nicotine biomarkers; both test results will be the basis for incentive payments. Asthma control will be evaluated using validated questionnaires and review of the participant's electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver aged greater than 18 years who is an active smoker.
* Child aged 2-12 years of age who meets clinical criteria for persistent asthma and has nicotine biomarker levels consistent with secondhand smoke exposure
* Designated social network member who is an active smoker
* Residence in Baltimore City

Exclusion Criteria:

* Child has current diagnosis of another major pulmonary disease or other significant medical co-morbidity
* Use of electronic cigarettes (e-cigarettes) by the adult-enrolled participants

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Pediatric secondhand smoke exposures | 6 months
  Monthly measurement of pediatric secondhand smoke exposures. Secondhand smoke exposures will be measured using salivary cotinine levels.

SECONDARY OUTCOMES:
Nicotine biomarkers | 6 months
  Monthly measurements of nicotine biomarkers to objectively assess tobacco usage. This will serve as the trigger for monthly financial incentives for those allocated to the intervention group.
Air nicotine | 6 months
  Home air nicotine levels will be measured to assess if tobacco-derived indoor air pollutant levels will decline with the intervention. Air nicotine levels will be acquired through passive air samplers and measured using gas chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep S Jassal, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jassal MS, Lewis-Land C, Thompson RE, Butz A. Randomised pilot trial of cash incentives for reducing paediatric asthmatic tobacco smoke exposures from maternal caregivers and members of their social network. Arch Dis Child. 2021 Apr;106(4):345-354. doi: 10.1136/archdischild-2019-318352. Epub 2020 Oct 1. PMID 33004310